CLINICAL TRIAL: NCT05018039
Title: A Mixed-methods Randomised Feasibility Trial Comparing a Collaborative Care Model With Standard Care in People With Musculoskeletal and Co-existing Mental Health Conditions.
Brief Title: Feasibility and Acceptability of Collaborative Care for People With Musculoskeletal and Mental Problems
Acronym: CCOPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Iva Hauptmannova, Head of Research Innovation Centre, Royal National Orthopaedic Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21.06
Record Dates: First submitted 2021-06-30; First posted 2021-08-24 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Mental Disorder; Musculoskeletal Diseases
Keywords: Collaborative Care Model; Case Manager; RCT; Feasibility; Mixed Methods
MeSH Terms: conditions — Mental Disorders; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative care model (Experimental): Collaborative care involves three professionals: a physical health care provider (physiotherapist or occupational therapist), a mental health care provider (psychologist or psychiatrist) and a case manager. The case manager will work closely with the patient to identify the mental health support necessary. This may involve appointments with a psychologist or psychiatrist as part of their musculoskeletal treatment.
  The case manager will define a treatment plan and organise appointments with the patients and monitor their progress using validated questionnaires, adjusting their mental or physical care support when required. This professional will also monitor patients' attendance and support managing their appointments and routinely update the clinical team on patient progress, and relaying information back to the clinical team. This model of care will work in parallel to the regular musculoskeletal appointments with the physiotherapist and/or occupational therapist (usual care).
  Interventions: Other: Collaborarive Care Model
- Usal Care (No Intervention): Current usual care within musculoskeletal outpatients involves an initial patient assessment by a physiotherapist or occupational therapist (or both) to determine the needs and goals of the patient in relation to their musculoskeletal condition. Clinicians also help to inform, educate, and empower patients to self-manage their rehabilitation where possible.
  Following this initial assessment, patients are provided with a plan of their therapy treatment. The therapist(s) progress patients exercise, as appropriate. Therapy is most often a 1:1 session but can also include group classes. Physical therapy involves exercise and education, while occupational therapy focuses on practical strategies to perform daily tasks.
  If the therapists feel that patients require additional support for their mental health problems, they can request this support via the General Practitioner or the hospital mental health services.

INTERVENTIONS:
Other: Collaborarive Care Model — Collaborative care involves three professionals: a physical health care provider (physiotherapist or occupational therapist), a mental health care provider and a case manager. The case manager will work closely with the patient to identify the mental health support necessary. This may involve appointments with a psychologist or psychiatrist as part of their musculoskeletal treatment.
  The case manager will define a treatment plan and organise appointments with the patients and monitor their progress using validated questionnaires, adjusting their mental or physical care support when required. This professional will also monitor patients' attendance and support managing their appointments and routinely update the clinical team on patient progress, and relaying information back to the clinical team. This model of care will work in parallel to the regular musculoskeletal appointments (usual care).
  Arms: Collaborative care model

SUMMARY:
This study aims to implement a feasibility Randomised Controlled Trial to support patients with musculoskeletal problems and a co-existing mental condition, which the intervention will be the implementation of a Collaborative Care Model.

In England, one in six adults suffers from a mental health condition, such as anxiety or depression. Despite these high numbers, mental health conditions are often unrecognised in physical healthcare settings, including patients with musculoskeletal (MSK) conditions. Patients with both a physical and mental health diagnosis are likely more difficult to treat in comparison to those with just a physical health condition.

The Collaborative Care Model offers an alternative way of improving musculoskeletal rehabilitation as it takes into consideration both physical and mental health needs. This model involves physical and mental healthcare professionals working together to better identify and manage people with both conditions. Patients are then further supported by a Case Manager who coordinates access to relevant professionals/services following an assessment of both physical and mental health needs.

The investigators propose a feasibility study to assess whether the collaborative care model is beneficial to orthopaedic patients in addressing both physical and mental health needs.

Patients over 18 years old, with an MSK condition attending therapy services at the Royal National Orthopaedic Hospital with a moderate to severe anxiety or depression score, may be eligible. Following informed consent, they will be randomly allocated to either treatment as usual or the intervention group (the collaborative care model with input from a Case Manager). All participants will participate for 6 months with a follow-up on months 3 and 6.

DETAILED DESCRIPTION:
Methodology:

The investigators will perform a single-center, mixed methods two-arm parallel-group Randomized Control trial (RCT), comparing the collaborative care intervention in patients with musculoskeletal (MSK) and co-existing mental conditions with usual care.

The study will be carried out at the Therapies Rehabilitation Outpatient setting, at the Royal National Orthopaedic Hospital NHS Trust, Stanmore, London. The duration of the study will be 12 months and the patient's participation will be for 6 months.

Patients will be approached by their attending physician in their routine outpatient clinic appointment regarding whether they would be interested in taking part in this study. As per routine care, this patient group complete PHQ-ADS in their outpatient appointment.

If the patient is interested in taking part and has a PHQ-ADS score of >20, they will be referred to the research team to further discuss participation. The study team will be introduced and available to discuss the study with potential participants. A written patient information sheet (PIS) will be provided. Patients will be given time to process the information should they be interested (a minimum of 24 hours), and consent will be obtained at their next routine appointment, once patients have read and understood the PIS.

Randomised Control Trial:

Following written informed consent, participants will be randomized in a 1:1 ratio (usual care: intervention) which will be undertaken via an online randomization software.

Sample:

It is proposed to recruit 40 patients in total, 20 randomized to each arm of the study. As the study is a feasibility trial, all analyses will be descriptive, with no hypothesis testing. As such no formal sample size calculation has been conducted.

All potentially eligible participants will be recruited through the direct clinical care team. Over 4,000 new patients are attending the therapies appointments annually and they need to complete the PHQ-ADS as a routine of their care.

Data collection:

Data will be collected through questionnaires administrated in clinical, telephone, or video calls according to participant preference and availability. At the eligibility assessment, the PHQ-ADS is collected as a routine of the outpatients setting.

Baseline data will be collected from participants on both arms, including demographic data (age, ethnicity, marital status, highest qualification level, employment status, type of musculoskeletal and mental conditions known and treatment), medical history and current medication using a tailored questionnaire.

The participant will also be asked to complete other quantitative measures at the baseline visit (approx. 50 minutes). This will include self-reported measures of depression, anxiety, pain, and quality of life. These questionnaires will also be completed on month 3 and 6 follow-ups, including any update on the current medication. Participants will stay in the study for a total of 6 months.

Interviews and Focus Group:

Once participant involvement in the study is complete to assess the acceptability of this model of care, participants from the intervention group will be invited to interviews, and health care professionals will be invited for a focus group. The interviews and focus groups will be optional.

Patient interviews will last for approximately 1 hour with some guided topics. The interview is planned to happen face-to-face at the RNOH. Nevertheless, due to COVID restrictions or participant preference, video or telephone interviews will also be available options. Interviews will avoid breaches of confidential material regarding participants' mental health conditions.

The focus group for staff will occur at the end of the RCT. There will be an estimated 6 to 10 members of staff in the focus group, and it will last for approximately 90 minutes. It will take place in RNOH and will be scheduled to suit staff availability. The trial aims to hold face-to-face focus groups but due to COVID restrictions, these focus groups will also be offered on an online platform. It is not expected for staff to attend more than one session, but the staff is welcome to attend another session if they have further feedback to contribute.

This data will give us a chance to understand the experience of being involved in the intervention group. The investigators would like to know the views, thoughts, and experiences of the participants; for example, their opinions on working with a Case Manager, potential advantages, and challenges.

Quantitative data analysis:

The primary analysis will estimate the number of potentially eligible participants, consent and overall uptake. The retention and adherence rates will be calculated in relation to the number of participants recruited. Standard deviations and confidence intervals of clinical outcomes will be calculated and used to determine which outcomes are most sensitive to change which will inform the sample size calculation for a future multi-centre RCT. The staff costs for the intervention group will be calculated using the National Cost index for the NHS.

A statistical analysis plan will be developed by the study statistician supported by SPSS software version 27.

Qualitative data analysis:

Focus groups and interviews will be transcribed in full (ipsis verbis) by an external company, checked for accuracy by a Principal Investigator and then imported into NVIVO version12 qualitative data analysis software, to aid management and indexing of data.

The analysis will begin shortly after data collection starts and framework analysis with Normalization Process Theory (NPT) will be used by the Principal Investigator (Jo). This type of analysis explains processes by which complex interventions become routinely embedded in health care practice. Transcripts from the participants and health care professionals will be analyzed separately. A subset of transcripts will be independently double coded by the other member of the research team and compared. Discrepancies will be discussed and resolved to achieve a coding consensus.

It is aimed to obtain a deeper understanding of the acceptability of the intervention, resources needed, and disclose potential barriers and facilitators from the participants' and health care professionals' points of view.

ELIGIBILITY:
Participants/ patients

Inclusion Criteria:

* Patients over 18 years old, with an MSK condition requiring a therapy outpatient appointment.
* Scoring ≥ 20 on the PHQ-ADS.
* Able to provide written informed consent and willing to participate
* Able and willing to complete questionnaires and study assessments

Exclusion Criteria:

* Patients who are already receiving treatment for a psychiatric condition from a specialist mental health service.
* Scoring < 20 on the PHQ-ADS.
* Lacking capacity to consent
* Unable or unwilling to complete questionnaires and study assessments
* Participating in other trials

Participants/ staff

Clinical staff involved in the treatment of the participants allocated to the intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants | 6 months
  Number of participants consented as a proportion of the number of patients eligible and invited.
Retention | 6 months
  Number of participants ending the trial as a proportion of the number of patients recruited.
Protocol adherence | 6 months
  Percentage of appointments attended as a proportion of booked appointments (%)

SECONDARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | pre-intervention, 3 months and 6 months
  From 0 (no anxiety and depression) to 45 (severe anxiety and depression).
  This assessment does not include units.
Resourcing | month 6
  Resources needed to implement the collaborative care model does not include measurements/units
  Usage of concomitant health services - Type of services and frequency of use in absolute numbers
  Implementation facilitators and barriers in the intervention arm - qualitative data that will collect via interviews and focus group
  Patient and staff acceptability of the intervention - qualitative data that will collect via interviews and focus group
  Cost of clinical staff involved on the intervention arm - thorough the number, type and duration of appointments performed by case manager, therapists, and mental health specialist
NPRS | pre-intervention, 3 months and 6 months
  From 0 to 10
  These assessments do not include units
Pain Disability Index (PDI) to assess pain | pre-intervention, 3 months and 6 months
  From No Disability 0 to Worst Disability 10
  These assessments do not include units
Quality of life validated Questionnaire EQ-5D | pre-intervention, 3 months and 6 months
  This scale is numbered from 0 to 100. 100 means the best health you can imagine. 0 means the worst health you can imagine.
  This assessment does not include units
Physical health quality assessment validated questionnaire (MSK-HQ) | pre-intervention, 3 months and 6 months
  To assess pain severity, physical function, work interference, social interference, sleep, fatigue, emotional health, physical activity, independence, understanding, confidence to self-manage and overall impact.
  The MSK-HQ total score is the sum of items 1-14 from 0 (worst impact) to 56 (no impact).
  This assessment does not include units
Global rating of change assessment validated questionnaire (GROC) | pre-intervention, 3 months and 6 months
  To assess self-perceived improvement
  From options a very great deal worse to a very great deal better.
  This assessment does not include units.

CONTACTS AND LOCATIONS:
Overall Officials: Parashar Ramanuj, MBBS, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust
Locations (2):
- United Kingdom (2):
  - Iva Hauptmannova, Stanmore, London
  - Royal National Orthopaedic NHS Trust, Brockley Hill, Stanmore, UK

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Teixeira MJC, Ahmed R, Tehrany R, Jaggi A, Ramanuj P. Collaborative care model versus usual care for the management of musculoskeletal and co-existing mental health conditions: a randomised feasibility mixed-methods study. BMJ Open. 2024 Feb 21;14(2):e079707. doi: 10.1136/bmjopen-2023-079707. PMID 38387980